CLINICAL TRIAL: NCT01215370
Title: Effect of Arginine-rich Dietary Protein on Postprandial Metabolism, Inflammation and Endothelial Function
Brief Title: Pea Protein and Postprandial Response (PEA)
Acronym: PEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Wageningen University (Division of Human Nutrition ), Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL3207808110 (Other: Medical Ethics Review Committee)
Record Dates: First submitted 2010-09-30; First posted 2010-10-06 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pea Proteins; Glutens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: High-fat shake with Pea protein — Shake containing 95 gram of fat, additive 30 gram pea protein
  Other Names: Experimental
Other: High-fat shake with Pea protein hydrolysate — Shake containing 95 gram of fat, additive 30 gram gluten protein hydrolysate
  Other Names: Experimental
Other: High-fat shake - Control — Shake containing 95 gram of fat, no protein additive
  Other Names: Control
Other: High-fat shake with Gluten protein — Shake containing 95 gram of fat, additive 30 gram gluten protein.
  Other Names: Experimental
Other: High-fat shake with Gluten protein hydrolysate — Shake containing 95 gram of fat, additive 30 gram gluten gluten hydrolysate
  Other Names: Experimental

SUMMARY:
The main objective is to investigate the postprandial effect of arginine-rich protein (i.e. pea-protein) on metabolic control, inflammation and endothelial function after a high-fat meal in subjects with characteristics of the metabolic syndrome.

DETAILED DESCRIPTION:
Arginine is potential interesting considering the metabolic syndrome. Studies so far indicated both long-term effects, as well as acute - postprandial - actions; especially when metabolism is already challenged, e.g. in diabetic patients or after a high-fat meal. If arginine-rich proteins are equally effective is not known. Therefore we are interested in the effect of (arginine rich) protein on postprandial (dys)metabolism, inflammation and endothelial function, within 6 hours after a meal.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* central obesity: waist circumference ≥94 cm

plus any one of the following four factors:

* raised triglyceride level: ≥1.7 mmol/L;
* reduced high-density lipoprotein (HDL) cholesterol: <1.03 mmol/L
* raised blood pressure: systolic blood pressure ≥130 mmHg or diastolic BP ≥85 mmHg or use of blood pressure lowering medication
* raised fasting plasma glucose ≥ 5.6 mmol/L

Additional inclusion criteria:

* age 45-70 years
* body weight should be stable for 3 months
* stable exercise habits during the last 6 months, and not participating in any vigorous exercise program

Exclusion Criteria:

* tobacco smoking
* (undiagnosed) diabetes - but not impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) as evaluated by an oral glucose tolerance test at screening
* active hearth disease, i.e. history of myocardial infarction or angina pectoris
* following, or have recently followed a (weight-loss) diet
* drug uses knowing to interfere with the objectives of the study
* oral corticosteroids, lipid-lowering drugs (statins)
* allergic to cow milk / dairy products or gluten
* vegetarians
* received inoculations within 2 months of starting or planned to during the study
* donated or intended to donate blood 2 months before till two months after the study
* abuse of drugs and/or alcohol
* participation in another biomedical study within 1 month before the first screening visit
* not agreeable to be informed about possible distorted blood values which could be found by screening

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Postprandial metabolic, inflammatory and endothelial response | up to 6 hours
  Metabolic: Plasma glucose, insulin and triglyceride levels (T= 0,1,2,3,4,5 and 6 hrs)
  Inflammatory: C-reactive protein (CRP), Plasminogen activator inhibitor-1 (PAI-1), Tumor necrosis factor-alpha (TNF-a), Interleukin-6 (IL-6), Inter-Cellular Adhesion Molecule-1 (ICAM-1) and Monocyte chemotactic protein-1 (MCP-1) (T=0, 2, 4 and 6 hrs).
  Endothelial function: Macro vascular regional arterial stiffness by Pulse Wave Analysis (PWA) (T=0, 3 and 6 hrs).

SECONDARY OUTCOMES:
Satiety markers and Oxidative stress | up to 6 hours
  Satiety: Glucagon-like peptide-1 (GLP-1) (T=0,2,4 and 6 hrs).
  Oxidative stress: Peripheral blood mononuclear cells (PBMC) (T=0,3 and 6 hrs).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mensink, Dr, Study Chair — Department Human Nutrition, Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands